CLINICAL TRIAL: NCT00187083
Title: A Study of Children With Refractory or Relapsed Acute Lymphoblastic Leukemia (ALLR16)
Brief Title: A Study of Children With Refractory or Relapsed ALL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Name/Official Title: Sima Jeha, MD / Principal Investigator, St. Jude Children's Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALLR16
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Leukemia; Acute Lymphoblastic Leukemia; Refractory Acute Lymphoblastic Leukemia; Relapsed Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — Topotecan; Dexamethasone; Vincristine; pegaspargase; asparaginase erwinia chrysanthemi recombinant; fludarabine; Methotrexate; Mercaptopurine; Idarubicin; Etoposide; Teniposide; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Native asparaginase
  Interventions: Drug: Topotecan, dexamethasone, vincristine; Drug: E. coli Asparaginase, PEG-L-asparaginase; Drug: erwinia asparaginase; Drug: fludarabine, methotrexate, mercaptopurine; Drug: idarubicin, etoposide, cytarbine, teniposide; Procedure: chemotherapy, intrathecal chemotherapy, steroid therapy
- 2 (Experimental): PEG-asparaginase
  Interventions: Drug: Topotecan, dexamethasone, vincristine; Drug: E. coli Asparaginase, PEG-L-asparaginase; Drug: erwinia asparaginase; Drug: fludarabine, methotrexate, mercaptopurine; Drug: idarubicin, etoposide, cytarbine, teniposide; Procedure: chemotherapy, intrathecal chemotherapy, steroid therapy

INTERVENTIONS:
Drug: Topotecan, dexamethasone, vincristine — See Detailed Description section for details of treatment interventions.
Drug: E. coli Asparaginase, PEG-L-asparaginase — See Detailed Description section for details of treatment interventions.
Drug: erwinia asparaginase — See Detailed Description section for details of treatment interventions.
Drug: fludarabine, methotrexate, mercaptopurine — See Detailed Description section for details of treatment interventions.
Drug: idarubicin, etoposide, cytarbine, teniposide — See Detailed Description section for details of treatment interventions.
Procedure: chemotherapy, intrathecal chemotherapy, steroid therapy — See Detailed Description section for details of treatment interventions.

SUMMARY:
The main purpose of this study is to find out which form of asparaginase (the native E. coli/Erwinia) or PEG-asparaginase) is more effective during induction treatment for children with acute lymphoblastic leukemia that has come back after treatment (relapsed) or is resistant to treatment (refractory)

DETAILED DESCRIPTION:
The present protocol will compare the biologic effects of PEG-asparaginase vs native-forms of asparaginase in a randomized trial using the same dosages and schedules used in the POG 9411 study. Comprehensive studies, including the measurement of antibodies and asparagine levels as well as the pharmacokinetics of L-asparaginase, will be performed. This protocol will also study the changes in topoisomerase I and topoisomerase II levels and the fractions of topoisomerase I/II translocations in malignant lymphoblasts after upfront window topotecan therapy, and correlate oncolytic response with these changes.

Secondary objectives include:

* To compare changes in asparagine levels 28 days after initiation of treatment with asparaginase between the two groups.
* To estimate the pharmacokinetics of L-asparaginase, compare the pharmacokinetics between the two groups of patients, and correlate the pharmacokinetics with the development of antibody to asparaginase and depletion of asparagine.
* To measure the pharmacokinetics and pharmacodynamics of topotecan in patients with recurrent acute lymphoblastic leukemia
* To determine whether the frequency of recombinogenesis in lymphocytes is increased during or after etoposide therapy relative to the pre-therapy level, and to explore whether etoposide pharmacokinetics are related to the Day 7 or post-therapy level of recombinogenesis.

Detailed Description of Treatment Plan

WINDOW Topotecan 2.4 mg/m2 ; IV over 30 min in 5 doses Days 1-5

STANDARD INDUCTION Dexamethasone 6 mg/m2/day orally Days 8-35 Vincristine 1.5 mg/m2 (max 2.0 mg) days 8, 15, 22, 29

RANDOMIZE E. coli asparaginase 10,000 U/m2/day IM (or Erwinia if previous allergy to E. coli) Days 8, 11, 13, 15, 18, 20, 22, 25, 27, 29, 32, 34

OR

PEG-Asparaginase 2500 U/m2/day IM Days 8, 15, 22, 29

ITHMA Days 8, 22, 36

CONSOLIDATION

Fludarabine: 15 mg/m2 IV over 30 min; days 1,2,3,4 Ara-C: 2 g/m2 IV days 1,2,3,4

Patients who achieve remission on R16 induction or consolidation may be eligible for either a matched sibling or a fully matched/one-antigen-mismatched unrelated donor transplant

For patients not undergoing bone marrow transplant:

SECONDARY CONSOLIDATION

VP 16: 50 mg/m2 PO qd for 14 days. Vincristine: 1.5 mg/m2 (max 2.0 mg) IV; days 1, 8. IT MHA day 1

CONTINUATION CHEMOTHERAPY

Cycle 1:

Cyclophosphamide 1 g/m2 IV on days 1 and 2 Vincristine 1.5 mg/m2 IV on day 1 (max 2.0 mg)

Cycle 2:

VP-16 50 mg/m2 day PO daily x 14 days Decadron 6 mg/m2 PO daily ) TID x 14 days Vincristine 1.5 mg/m2 IV (max 2 mg) on days 1 and 8.

Cycle 3:

HD MTX 5 gm/m2 continuous infusion over 24 hrs E. coli Asparaginase 10,000 U/m2/dose IM qod x3 or PEG Asparaginase 2500 U/m2/dose IM x 1 (maintain same randomization for Asparaginase preparation as during induction)

Cycle 4:

High Dose Ara-C 2 g/m2/dose IV over 2 hrs q 12 hrs x 3 doses.[Total dose 6 gm/m2] Idarubicin 12 mg/m2 IV over 30 min X 1 [after completion of first dose of Ara-C] IT MHA on day 1 prior to the HDARA-C (dose of ITMHA is age adjusted as outlined in section 7.3)

STANDARD CONTINUATION CHEMOTHERAPY

Patients will receive 4-week rotational cycles of chemotherapy with the following pairs of drugs for total treatment duration of 17 months.

Week #1 Cyclophosphamide (300 mg/m2 IV) + VCR (1.5 mg/m2 IV; max 2 mg). Week #2 VM26 (200 mg/m2 IV) + Ara C (300 mg/m2 IV). Week #3 MTX (MTX should be given IM or as a 2 hr IV infusion if the patient has had previous cranial iradiation) (40 mg/m2 IV/IM) + 6 MP (75 mg/m2 PO q HS x 7) Week #4 MTX (MTX should be given IM or as a 2 hr IV infusion if the patient has had previous cranial irradiation)(40 mg/m2 IV/IM) + 6 MP (75 mg/m2 PO q HS x 7)

IT MHA: Given every 8 weeks throughout standard continuation chemotherapy for patients with CNS 1 status Given every 4 weeks for patients with CNS 2/3 status who will receive CSI at the end of chemotherapy

ELIGIBILITY:
Inclusion Criteria

For patients treated on frontline protocols at St. Jude:

* ALL in isolated bone marrow relapse, or combined marrow and extramedullary relapse, during or after treatment with multi-agent chemotherapy (TOTAL XI, XII, XIIIA, XIIIB), or isolated extramedullary relapse after treatment on TOTXII.
* Patients with recurrent T-Cell non-Hodgkin's lymphoma who relapse in the bone marrow with >25% blasts

For patients not treated on front-line St. Jude protocols:

• ALL in isolated bone marrow relapse, or isolated extramedullary relapse, or combined marrow and extramedullary relapse.

All patients:

* First relapse after receiving primary therapy or during primary therapy
* Life expectance of at least 8 weeks
* ECOG score 0-2 Exclusion criteria
* Life expectancy < 8 weeks

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 1997-02; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
To compare in a randomized trial the depletion of asparagine in patients who receive the native form of asparaginase or PEG-asparaginase during induction therapy. | December 2003

CONTACTS AND LOCATIONS:
Overall Officials: Sima Jeha, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: Related Info — http://www.stjude.org